CLINICAL TRIAL: NCT05024682
Title: Pulsed Radiofrequency Versus Pulse Dose Pulsed Radiofrequency of the Pudendal Nerve in Patients With Pudendal Neuralgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Saeid Metwaly Abouelyazid Elsawy, DR, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: wx1569
Record Dates: First submitted 2021-08-22; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- conventional pulsed radiofrequency (Experimental)
  Interventions: Device: conventional pulsed radiofrequency
- pulse dosed pulsed radiofrequency (Experimental)
  Interventions: Device: pulse dosed pulsed radiofrequency

INTERVENTIONS:
Device: conventional pulsed radiofrequency — After connecting the electrode and the PRF needle, the interventionist determined whether the pudendal nerve innervation produced paresthesia in the sensory stimulation test with a frequency of 50 Hz, pulse width of 1 ms and a voltage of 0.3-0.5 V. Thereafter, the radiofrequency ablation therapy was performed in 42°C, 120 seconds pulse mode which consisted of four cycles (8 minutes)
  Arms: conventional pulsed radiofrequency
Device: pulse dosed pulsed radiofrequency — After connecting the electrode and the PRF needle, the interventionist determined whether the pudendal nerve innervation produced paresthesia in the sensory stimulation test with a frequency of 50 Hz, pulse width of 1 ms and a voltage of 0.3-0.5 V. Thereafter, the radiofrequency ablation therapy was performed in 42°C, 240 seconds pulse dose mode which consisted of two cycles (8 minutes).
  Arms: pulse dosed pulsed radiofrequency

SUMMARY:
The relatively complex anatomical structure of the pelvis has been a focus of study in the medical field. The diagnosis of the causes of chronic pelvic pain is usually a complicated process.

Pudendal neuralgia is a syndrome that is characterized by pelvic pain, including bowel, bladder regional pain or discomfort, sexual dysfunction, severe burning sensations and needle-like pain, which are aggravated when seated and relieved after standing. pudendal neuralgias are induced by pudendal nerve damage The mechanism of PRF has been studied repeatedly. It has been verified that PRF has definite safe treatment range, but during the PRF treatment, the tissue surrounding the electrode may have some degree of change and so it is difficult to assess any actual damage.7 Based on electric field intensity, PRF can actually produce tissue changes observable as in vitro changes to ultrastructure in early-phase histologic study. These biological changes were converted to biological effect to alleviate neuropathic pain in animal models.

ELIGIBILITY:
Inclusion Criteria:

* pain located in the pudendal nerve distribution area
* pain intensity increases in the sitting position;
* no nocturnal pain symptoms;
* pain with no objective sensory impairment
* pain is relieved by diagnostic pudendal
* the pain symptom is associated with sexual dysfunction, with the elimination of obstetrical and gynaecologic, urological and anorectal diseases in the related departments and absence of any physical and mental disorders;
* treatment by other departments is invalid;
* patients should be older than 18 years
* patients should be able to sign an informed consent form

Exclusion Criteria:

* patients have simple tailbone, gluteus muscle or lower abdominal pain, or only paroxysmal pain, or only pruritic symptoms, and/or have imaging anomalies that may explain the symptoms;
* female patients who are pregnant;
* patients who take anticoagulant drugs or have any coagulation disorder;
* patients who are unable to complete the questionnaire;
* patients with pain, which is caused by malignant or autoimmune diseases and
* patients who are hypersensitive to metals.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-03 (Estimated); Primary Completion 2023-01-03 (Estimated); Study Completion 2023-02-03 (Estimated)

PRIMARY OUTCOMES:
visual analogue score | 3 months
  The VAS score was used that has 0-10 points. The 0 point represents the painless state and a score from 1 to 3 points represents mild pain, from 4 to 6 points represents moderate pain and from 7 to 10 points represents severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Saeid Metwaly Elsawy, Asyut, Egypt